CLINICAL TRIAL: NCT01031472
Title: A Single-center, Randomized, Two Part, Open-label, Crossover Study to Assess the Relative Bioavailability and Food Effect of New Formulations of GSK2248761 in Healthy Adult Subjects
Brief Title: A Study to Assess Relative Bioavailability and Food Effect of New Formulations of GSK2248761
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113391
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: HIV, relative bioavailability, food effect, GSK2248761, healthy subjects; HIV Seronegativity
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will be randomized in a three way crossover design to either a single dose of GSK2248761 100mg Gelucire capsule administered with food and a single dose of 100mg of formulation 1 or a single dose of 100mg of formulation 3 administered in the fed and fasted state
  Interventions: Drug: GSK2248761 formulation 1; Drug: GSK2248761 reference formulation; Drug: GSK2248761 formulation 3
- Part B (Experimental): A total of twelve subjects who complete Part A will participate in Part B. Subjects from Part A will be asked to participate on a first come first serve basis until there are 12 subjects, at which time enrolment to Part B will be closed. Part B will be a 2 way cross over study design. Subjects will be randomized to one of a single dose of GSK2248761 100mg Formulation 2 or 4 (based on the evaluation of Part A data) administered with food or in the fasted state. Subjects in Part B will not receive the reference formulation since they previously received this in Part A
  Interventions: Drug: GSK2248761 formulation 2 or 4

INTERVENTIONS:
Drug: GSK2248761 formulation 1 — 100mg GSK2248761 formulation 1- fasted 100mg GSK2248761 formulation 1 - with food (moderate fat meal)
  Arms: Part A
Drug: GSK2248761 reference formulation — GSK2248761 100mg Gelucire reference capsule with food
  Arms: Part A
Drug: GSK2248761 formulation 3 — 100mg GSK2248761 formulation 3 fasted 100mg GSK2248761 formulation 3 with food (moderate fat meal)
  Arms: Part A
Drug: GSK2248761 formulation 2 or 4 — 100mg GSK2248761 formulation 2 or 4 - fasted 100mg GSK2248761 formulation 2 or 4 - with food (moderate fat meal)
  Arms: Part B

SUMMARY:
This is a single-center, randomized, two part, open-label, crossover study in healthy adult subjects to assess the effect of up to three formulations on the relative bioavailability of GSK2248761 100mg administered with and without food. Part A will evaluate two new formulations compared to the current formulation. Part B will evaluate one additional formulation if the bioavailability of the two formulations in Part A do not meet pre-specified criteria. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-10 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECGs.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 MlU/ml is confirmatory.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* The subject has received GSK2248761 in a previous clinical trial.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period. Note: this does not include plasma donation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects at Screening and predose Day 1.
* Cardiac conduction abnormalities on a single 12-lead ECG at screening or predose Day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2010-03-11 (Actual); Study Completion 2010-03-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve zero to infinity of plasma GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of AUC (0-inf) of GSK2248761.
AUC from time zero to end of dosing interval AUC (0-tau) | Up to 5 weeks
  Plasma samples will be collected for the analysis AUC (0-tau) of GSK2248761.
Maximum concentration (Cmax) of GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of Cmax of GSK2248761.

SECONDARY OUTCOMES:
Terminal half life (t1/2) of GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of t1/2 of GSK2248761.
Lag time before observation of drug concentration (tlag) of GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of tlag of GSK2248761.
Time to Cmax of GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of Tmax of GSK2248761.
Percentage of AUC obtained by extrapolation (%AUCex) for GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of %AUCex for GSK2248761.
Apparent clearance following oral dosing (CL/F) for GSK2248761 | Up to 5 weeks
  Plasma samples will be collected for the analysis of CL/F for GSK2248761.
Number of participants with seious adverse events (SAEs) and non-serious adverse events (non-SAEs) | Up to 5 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement.
Number of participants with concurrent medication | Up to 5 weeks
  Number of participants with concurrent medication will be summarized.
Number of participants with abnormal clinical laboratory parameters | Up to 5 weeks
  Blood samples will be collected for the analysis of clinical laboratory parameters.
Number of participants with abnormal electrocardiogram (ECG) values | Up to 5 weeks
  12-lead ECG will be obtained using an ECG machine. Participants will be in supine or a semi-recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs are recorded.
Number of participants with abnormal vital signs | Up to 5 weeks
  Vital signs will be measured at indicated time points in semi-supine position after 5 minutes rest.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 113391 can be found on the ViiV Clinical Study Register. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=113391&attachmentIdentifier=98949e52-f1b5-4212-95ad-8ba8bebe8466&fileName=44f6043f-cd36-4fde-9b4a-3e28712ecce0.pdf&versionIdentifier=